CLINICAL TRIAL: NCT01451047
Title: A Phase 2 Randomized Study to Evaluate and Compare the Efficacy of Injections of ex Vivo Expanded Cultured Occipital Autologous Dermal and Epidermal Cells vs. Dermal Cells Into the Balding Scalp of Subjects With Hair Loss
Brief Title: A Study to Evaluate and Compare Injections of Autologous Dermal and Epidermal Cells Into the Balding Scalp of Subjects With Hair Loss (CA-0002012)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aderans Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CA-0002012
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Androgenetic Alopecia; Male Pattern Baldness; Female Pattern Baldness
Keywords: Androgenetic Alopecia; Male Pattern Baldness; Female Pattern Baldness; Hair Loss; Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Autologous cultured dermal and epidermal cells — A piece of occipital scalp is taken from the subject. The epidermal and dermal cells from this tissue are expanded in culture. The cells are then harvested and, for certain types of product, combined. These cells are then injected into the balding area of the scalp of the original subject.

SUMMARY:
To evaluate the ability of injections of Ji Gami(TM) and Ji Gami(TM) DO to induce hair growth in male and female subjects with hair loss

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers 18 to 65 years old, inclusive
* Hair loss consistent with ≥ Grade III-Vertex, IV, VA, V, and VI, based on Norwood-Hamilton Scale providing there is bridging of hair in the anterior edge of the vertex circle.
* Have no clinically significant disease or abnormal laboratory results taken at the screening visit.

Exclusion Criteria:

* Known sensitivity to DMEM/F-12 or any component of the study material.
* Known hypersensitivity to clindamycin hydrochloride, amphotericin B or streptomycin sulfate.
* Subjects who have used minoxidil, or any oral or topical medication including over the counter and herbal medications for the treatment of hair loss within 6 months of study screening, or finasteride or dutasteride within 12 months of study screening.
* A history of drug or alcohol abuse within 1 year of study enrollment.
* Clinically significant medical or psychiatric illness currently or within 30 days of study screening as determined by the investigator.
* Any clinically significant abnormal laboratory parameters.
* A positive result at screening for human immunodeficiency virus (HIV 1 or 2), Hepatitis B or C, HTLV I/II.
* Dermatologic condition in donation and/or study areas.
* Prior surgery in the treatment area.
* Insufficient hair or scarring in the donor area that might impact cell growth.
* Any disease or condition (medical or surgical) that, in the opinion of the investigator, might compromise hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system function; or any condition that would place the subject at increased risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hair number | 51 weeks post-injection
Change from baseline in hair width | 51 weeks post-injection
Time course of any treatment benefit | 51 weeks post-injection

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Atlanta, Georgia
  - Chicago, Illinois
  - Chevy Chase, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Raleigh, North Carolina
  - Houston, Texas